CLINICAL TRIAL: NCT00390702
Title: International Multicentre Clinical Device Investigation on Safety and Effectiveness of the Nit-Occlud® Lê VSD Spiral Coil System for VSD Occlusion Developed by Pfm AG, Cologne
Brief Title: Safety and Effectiveness of the Nit-Occlud® Lê VSD Spiral Coil System
Acronym: pfm-01/2005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: pfm medical gmbh (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pfm 01/2005
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Heart Septal Defects, Ventricular
Keywords: Ventricular septal defect; VSD
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VSD occluder (Experimental): transcatheter implantation of a VSD occluder (Nitinol coil)
  Interventions: Device: transcatheter implantation of a VSD occluder (Nitinol coil)

INTERVENTIONS:
Device: transcatheter implantation of a VSD occluder (Nitinol coil) — transcatheter implantation, by first performing a arterial-venous loop through the defect
  Other Names: Nit-Occlud® Lê VSD Occluder

SUMMARY:
The Ventricular septal defect (VSD) is the most common of all congenital cardiac malformations. By modifying the Nit-Occlud® PDA Device the Nit-Occlud® Lê VSD Spiral System was designed. as a percutaneous, transcatheter device for occlusion of (peri)membranous and muscular ventricular septum defects (VSD) with a spiral coil. In this clinical investigation feasibility, safety and performance of the new cardiac occluder will be evaluated in accordance with European and US regulations. The study data will be compared to performance criteria for VSD, which are deduced analogue to the published specific Objective Performance Criteria (OPCs) for PDAs. The first part of the study has been performed in three clinical centres in Germany. For the second part in April 2009 four additional clinical centres in Germany, Israel, Italy and Spain were included.

ELIGIBILITY:
Inclusion Criteria:

* VSD must be diagnosed by acknowledged methods, like echocardiography
* Signs of left ventricular volume overload are present (left ventricle or left atrium diameters 2 standard deviations greater than normal) and/or measured by catheterisation : Qp/Qs > 1.5
* Pulmonary vascular resistance is less than 4 Wood units
* The patient is older than 24 months
* The VSD has a perimembranous or muscular location.
* A distance between the rim of the VSD and the aortic annulus of at least 3.0 mm (as measured on the 2-D echocardiography - apical 5-chamber view)
* The minimal diameter (size) of the VSD is less than 8.0 mm (as measured on the 2-D echocardiography - apical 5-chamber view)
* Patient must agree to fully participate in the clinical trial and give informed consent in writing. If the patient is without legal ability additionally the person of legal responsibility must agree and s/he must give the informed consent in writing

Exclusion Criteria:

Pathological or physical condition precluding the implantation of a Nit-Occlud® Lê VSD coil, such as :

* perimembranous VSD with no evidence of circular aneurysm formation
* Associated cardiac anomalies requiring surgery (greater than mild aortic insufficiency; such as aortic valve prolapse)
* Active endocarditis or other type of sepsis or other active infection at time of implantation
* Thrombus at or near the intended site of implantation
* Thrombus in the vessels through which access to the VSD is gained (unless the patient is protected with an embolic protection device such as a vena cava filter)
* Vessels through which access to the VSD is gained can not accommodate a 7 F sheath
* Potential steric (3-dimensional) interference of the occluder with intracardiac or intravascular structures (like valves)
* History of blood disorder (coagulopathy, tendency towards haemolysis)
* History of hypersensitivity to contrast medium or Nitinol
* AV-block II° or III°, atrial fibrillation, or atrial flutter
* End stage cardiac disease, irreversible major organ failure, or terminal cancer
* HIV infection
* Cerebrovascular disease or neurological deterioration
* Emergency cardiologic intervention
* Patient*) is not able to fully participate in this study including all follow-ups (e.g. for mental or geographical reasons, or patient is intravenous drug user or has strong potential for non-compliance to medical regimes)
* Patient, respectively the person of legal responsibility, is mentally unable to understand the nature, aims, or possible consequences of the clinical investigation
* Pregnant or breast-feeding women
* Patient did participate in another clinical investigation during the last 3 months
* Patient or the person of responsibility has revoked the consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
a set of Performance Criteria (PC) deduced for VSD analogue to the set of Objective Performance Criteria (OPC) of the 'Multiorganization Advisory Panel to FDA for Pediatric Cardiovascular Devices' for PDAs | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meinertz, Prof Dr med, Principal Investigator — University Hospital Hamburg Eppendorf, Germany
Locations (6):
- Germany (5):
  - Dept. Congem.Heart Defects, Deutsches Herzzentrum, Berlin
  - Cardio-Vascular Centre, Sankt Kathrinen, Frankfurt
  - Univ.Klinikum, Zentrum fuer Kinderheilkunde, Giessen
  - Dept. Paediatric Cardiology, Univ. Hospital Hamburg, Hamburg
  - Dept. Paediatric Cardiology, Univ. Clinic Grosshadern, Munich
- Meyer Children's Hospital, Rambam Med. Center, Haifa, Israel